CLINICAL TRIAL: NCT03879876
Title: A Phase I/II Study Evaluating the Safety and the Efficacy of Human T Lymphoid Progenitor (HTLP) Injection to Accelerate Immune Reconstitution After Partially HLA Compatible Allogeneic Hematopoietic Stem Cell Transplantation in SCID Patients
Brief Title: Safety and Efficacy Study of Human T Lymphoid Progenitor (HTLP) Injection After Partially HLA Compatible Allogeneic Hematopoietic Stem Cell Transplantation in SCID Patients
Acronym: HTLP Necker
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150949J; 2018-001029-14 (EudraCT Number)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Patients; Any Type of Severe Combined Immunodeficiency (SCID); Partial HLA Incompatible Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: SCID; hematopoietic stem cell transplantation; Human T Lymphoid Progenitor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human T Lymphoid Progenitor (HTLP) injection (Experimental): Human T Lymphoid Progenitor cells (HTLPs) obtained after a brief period of ex vivo culture in the presence of the fusion protein DL-4, Retronectin® and a combination of cytokines
  Interventions: Drug: Human T Lymphoid Progenitor (HTLP) injection

INTERVENTIONS:
Drug: Human T Lymphoid Progenitor (HTLP) injection — Injection of progenitors derived from HTLP culture at Day 8-Day 12 after partially HLA compatible allogeneic hematopoietic stem cell transplantation in SCID patients (Day7 of culture)

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of Human T Lymphoid Progenitor (HTLP) injection to accelerate immune reconstitution after partially HLA compatible allogeneic hematopoietic stem cell transplantation in SCID patients.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients affected by any type of SCID confirmed by clinical, immunological and/or molecular diagnosis and eligible for an allogeneic HSCT
* Absence of a matched sibling donor or a matched unrelated donor (MUD) 10/10
* Clinical conditions incompatible with the search of a MUD
* Written, informed consent of parents/ legal representative (child)
* Age ≤ 2 years at the time of screening
* No prior therapy with allogeneic stem cell transplantation
* No treatment with another investigational drug within one month before inclusion
* Patient affiliated to social security

Exclusion Criteria:

* Presence of an HLA genoidentical donor
* Absence of written parental consent
* Treatment with another investigational drug within one month before inclusion
* Positive for HIV infection by genome PCR
* Contra-indication to allogeneic transplantation or conditioning therapy (except SCID patients with DNA repair deficiency)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-09-03 (Estimated); Study Completion 2025-06-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 3 months post-transplant
  to evaluate the procedure safety
reconstitution of the CD3+ TCRαβ+ cell compartment | Month 3
  determined by the presence of ≥ 300/µL total, circulating CD3+ TCRαβ+ T cells to evaluate the efficacy

SECONDARY OUTCOMES:
Time course of reconstitution of the different T cell subpopulations | Month 3, month 6, month 12
  time necessary to reach a normal number of naïve CD4+ and CD8+ T cells
presence of recent thymic emigrants | Month 3, month 6, month 12
  To evaluate the active thymopoiesis
T-cell receptor excision circles (TREC ) number in peripheral blood | Month 3, month 6, month 12
  To evaluate the active thymopoiesis
TCR rearrangements | Month 3, month 6, month 12
  By NGS analysis
B-cell reconstitution | Month 6, month 12
  number and phenotype for naïve IgD+CD27-, marginal zone IgD+CD27+, switched memory IgD-CD27+, and IgD-CD27- cells
Immunoglobulin (Ig) levels | Month 6, month 12
NK cell numbers | Month 6, month 12
Cumulative incidence of infections | 12 months post-transplant
Cumulative incidence of acute and chronic episodes of graft versus host disease (GVHD) | 24 months post-transplant
Overall survival | 2 years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ANDRE, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Despina MOSHOUS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris and Université Paris Descartes
Locations (1):
- Unité d'Immunologie Hématologie Rhumatologie Pédiatrique (UIHR),, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No